CLINICAL TRIAL: NCT04539795
Title: A Phase Ib/II, Single Center, Placebo-Controlled, Randomized, Blinded Study in Adult Patients (> 18 Years) With COVID-19 Respiratory Disease, to Evaluate, Safety, Tolerability and Mechanistic Effect of Alvelestat on Top of Standard of Care (COSTA)
Brief Title: COVID-19 Study of Safety and Tolerability of Alvelestat
Acronym: COSTA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mereo BioPharma (Industry)
Responsible Party: Principal Investigator, James Michael Wells, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300005845
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo oral tablet (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Alvelestat oral tablet - dose 1 (Active Comparator): MPH966
  Interventions: Drug: Alvelestat
- Alvelestat oral tablet - dose 2 (Active Comparator): MPH966
  Interventions: Drug: Alvelestat
- Alvelestat oral tablet - dose 3 (Active Comparator): MPH966
  Interventions: Drug: Alvelestat

INTERVENTIONS:
Drug: Alvelestat — oral tablet
  Other Names: MPH966
  Arms: Alvelestat oral tablet - dose 1; Alvelestat oral tablet - dose 2; Alvelestat oral tablet - dose 3
Drug: Placebo — oral tablet
  Arms: Placebo oral tablet

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics (PK), and explore the mechanistic and clinical effect of alvelestat (an oral neutrophil elastase inhibitor) orally twice per day for 10 days added to standard of care in adult patients (≥18 years) with COVID-19 respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age ≥18 years
* Proven SARS-Cov-2 infection (confirmed by PCR from a nasopharyngeal or lower respiratory tract sample)
* A score of Grade 3 to 5 on the WHO 9-point Ordinal Scale
* Male participants must agree to use a highly effective contraception during the treatment period and for at least 4 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants are eligible to participate if not pregnant; not breastfeeding; and at least one of the following conditions is met:

Not a woman of childbearing potential OR A woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment phase and for at least 4 days after the last dose of study medication - Capable of giving signed informed consent which includes a commitment to comply with the requirements and restrictions listed in the informed consent form (ICF) and within this protocol.

Exclusion Criteria:

* Patients who have previously had a score of 6 or 7 on the WHO 9-point Ordinal Scale
* Patients who require support with invasive mechanical ventilation at the time of inclusion, or expected to be required within 24 hours of randomization
* Alanine aminotransferase (ALT) OR aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) OR Total Bilirubin > ULN. In patients with a documented history of Gilbert's Syndrome AND baseline total bilirubin elevation consistent with an exacerbation of Gilbert's Syndrome (i.e. no other cause of total bilirubin elevation), subjects may enroll if total bilirubin is < 5x ULN.
* Diagnosis of liver cirrhosis, esophageal varices, ascites or hepatic encephalopathy
* Chronic liver diseases such as autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, Wilson's disease, haemochromatosis
* Significant renal disease or infection (as determined by the Investigator) including stage 4 chronic kidney disease or estimated glomerular filtration rate <60mL/min
* Absolute neutrophil count ≤ 1000/µL at screening
* Myocardial infarction, transient ischemic attack or stroke within 3 months prior to the first dose
* Current unstable angina or congestive heart failure (New York Heart Association III/IV)
* Screening 12-lead EKG with a measurable QTc interval according to Fridericia correction (QTcF) >450 ms
* Anticipated transfer to another hospital that is not the study center within 24 hours
* Allergy to study medication or excipients
* Inability to swallow tablets
* Other documented comorbidities or laboratory abnormalities that in the opinion of the Investigator could affect the outcome of the study assessments, participant safety, or ability of the participant to comply with the requirements of the protocol
* Any patient whose interests are not best served by study participation, as determined by the Investigator

Excluded Prior/Concomitant Therapy

* Requirement for medications mainly metabolized by CYP2C9 and with narrow therapeutic index (eg, warfarin, phenytoin) is prohibited unless therapeutic monitoring available for duration of alvelestat dosing
* Medicines that are potent CYP3A4 inhibitors including (but are not limited to) clarithromycin, diltiazem, erythromycin, itraconazole, ketoconazole, ritonavir, verapamil and potent inducers including but not limited to phenobarbital, phenytoin and rifampicin, will be exclusionary
* Requirement for medications substantially reliant on OATP1B1 for metabolism where discontinuation during study drug administration is not possible or where fluctuations in levels are considered clinically important (as per investigator judgement) and cannot be clinically monitored (e.g., statins, valsartan, olmesartan, enalapril, repaglinide)

Excluded Prior/Concurrent Clinical Study Experience

- Participation in any clinical investigation using investigational treatments within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the initial dosing (or longer if required by local regulations) is prohibited. Use of remdesivir (Veklury) under the conditions of the authorization for emergency use in the US, and per manufacturer's instructions, is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Wells, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Alvelestat Oral Tablet: MPH966
  Alvelestat: oral tablet
Period: Overall Study
Arm/Group | Placebo Oral Tablet | Alvelestat Oral Tablet
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: placebo
  Placebo: oral tablet
- Alvelestat: MPH966
  Alvelestat: oral tablet
- Total: Total of all reporting groups
Arm/Group | Placebo | Alvelestat | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (14.3) | 42 (23.9) | 47.8 (20.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Numbers and % of Subjects Who Experience at Least 1 Treatment-emergent Adverse Event
Description: Safety Outcome Assessment
Time Frame: to day 60
Measure: Count of Participants; unit: Participants
Groups:
- Alvelestat: Alvelestat
Arm/Group | Placebo | Alvelestat
Number analyzed (Participants) | 7 | 8
Participants | 3 | 5

2. Secondary Outcome: Effect of Alvelestat on Blood Pharmacodynamic Biomarkers of NETosis
Description: Change in blood markers of NETosis
Time Frame: Randomization through Day 10 or hospital discharge, whichever was shorter.
Measure: Mean (Standard Deviation); unit: log2(ng/ml)
Groups:
- Placebo: Placebo
Arm/Group | Placebo | Alvelestat
Number analyzed (Participants) | 7 | 8
log2(ng/ml)
  Cell-free DNA | -1.35 (2.66) | 0.16 (1.38)
  Citrullinated histone H3 | -.43 (1.94) | .73 (1.36)
  MPO-DNA | -.45 (1.01) | .53 (.48)
  MPO | -.39 (2.19) | .01 (1.04)

3. Secondary Outcome: Effect of Alvelestat on Blood Pharmacodynamic Biomarkers of Inflammation
Description: Change in blood markers of inflammation
Time Frame: Randomization through Day 10 or hospital discharge, whichever was shorter.
Measure: Mean (Standard Deviation); unit: log2(pg/ml)
Arm/Group | Placebo | Alvelestat
Number analyzed (Participants) | 7 | 8
log2(pg/ml)
  IL-1b | -1.37 (1.63) | 0.06 (1.14)
  IL-6 | 0.14 (2.37) | -1.61 (2.16)
  IL-8 | 0.56 (1.05) | -0.45 (0.76)
  TNFa | 0.61 (0.90) | -0.19 (0.58)

4. Secondary Outcome: Effect of Alvelestat on Blood Pharmacodynamic Biomarkers of D-dimer
Description: Change in blood markers of d-dimer
Time Frame: Randomization through Day 10 or hospital discharge, whichever was shorter.
Measure: Mean (Standard Deviation); unit: log2(ng/ml)
Arm/Group | Placebo | Alvelestat
Number analyzed (Participants) | 7 | 8
log2(ng/ml) | -0.08 (0.90) | -1.92 (2.89)

5. Secondary Outcome: Effect of Alvelestat on Blood Pharmacodynamic Biomarkers of Desmosine
Description: Change in blood markers of desmosine
Time Frame: Randomization through Day 10 or hospital discharge, whichever was shorter.
Measure: Mean (Standard Deviation); unit: log2(ng/ml)
Arm/Group | Placebo | Alvelestat
Number analyzed (Participants) | 7 | 8
log2(ng/ml) | -0.04 (1.14) | 0.54 (0.67)

6. Secondary Outcome: Mortality Rate
Time Frame: to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alvelestat
Number analyzed (Participants) | 7 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Placebo | Alvelestat
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/8
Other Adverse Events (participants affected / at risk) | 4/7 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Alvelestat (N=8)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) — Hospital readmission for worsening acute hypoxemic respiratory failure related to pneumonia due to COVID-19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Alvelestat (N=8)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT04539795/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT04539795/SAP_001.pdf